CLINICAL TRIAL: NCT02262676
Title: Observational and Cross-sectional Study to Assess the Sociodemographic and Clinical Characteristics of Patients Treated With RIVAROXABAN in the Context of Routine Clinical Practice of Spanish Haematologists, Cardiologists and Internists (HEROIC Study)
Brief Title: Observational Study to Assess Sociodemographic and Clinical Features of Patients Treated With Rivaroxaban in Routine Clinical Practice of Hematologists, Cardiologists and Internists of Spain
Acronym: HEROIC
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 17671
Record Dates: First submitted 2014-10-09; First posted 2014-10-13 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Atrial Fibrillation
Keywords: Stroke prevention on Atrial Fibrillation; Prevention and Control; Stroke
MeSH Terms: conditions — Atrial Fibrillation; Stroke | interventions — Rivaroxaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Rivaroxaban: Patients with Atrial fibrillation treated with Rivaroxaban
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto, BAY59-7939) — Patients treated by Physicians under approved local prescriptions

SUMMARY:
Depict demographic and clinical features of patients with atrial fibrillation treated with rivaroxaban to prevent stroke and pulmonary embolism in routine clinical practice

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years
* Patients with atrial fibrillation
* Patients in treatment with rivaroxaban for stroke prevention in atrial fibrillation at least 3 months previous to inclusion period in study

Exclusion Criteria:

* Patients in treatment after start of study
* Patients treated with other anticoagulant treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients taking rivaroxaban for stroke prevention in atrial fibrillation attending consults of hematology, cardiology and internal medicine
Sampling Method: Non-Probability Sample
Enrollment: 2251 (Actual)
Dates: Start 2014-10; Primary Completion 2015-02 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Demographic Data | At recruitment visit
Medical History | At recruitment visit

SECONDARY OUTCOMES:
Assess regional differences among the different Spanish autonomous communities on the management of patients with rivaroxaban treatment during the routine clinical practice | At recruitment visit
  By use of Informe de Posicionamiento Terapéutico (Spanish Questionnaire)
Adherence to rivaroxaban treatment | At recruitment visit
  By use of Morisky-Green questionnaire
Assess the satisfaction of rivaroxaban treatment | At recruitment visit
  By use of Anti-Clot Treatment Scale (ACTS) questionnaire
Assess the quality of life in patients | At recruitment visit
  By use of Short-Form 12 Health Survey,version 2 (SF12v2) questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Spain